CLINICAL TRIAL: NCT04270994
Title: Misoprotol as a Treatment for Endometrial Polyps in Infertile Patients
Brief Title: Misoprostol as a Treatment for Endometrial Polyps in Infertile Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Henry Aristoteles Mate-Sánez (Individual)
Responsible Party: Sponsor-Investigator, Henry Aristoteles Mate-Sánez, Principal Investigator, Mateo-Sánez, Henry A.
Organization: Mateo-Sánez, Henry A. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSP_2016
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Endometrial Polyps in Infertile Patients
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Misoprostol (Experimental)
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
Endometrial polyps are one of the main causes of infertility in women. In this work we propose an alternative, effective, economical and safe treatment: the use of misoprostol

DETAILED DESCRIPTION:
The prevalence of uterine polyps has been estimated in the general population at 10-15%, while in infertile patients it ranges from 6-32%. Its etiology is considered as multifactorial. Polyps induce a local inflammatory response in the endometrial cavity, causing infertility. The treatment of choice considered "gold standard" is the excision by hysteroscopy, however, improvement has been shown in patients with conservative management due to the regression rate of 27%. There are no recommended drugs to provide a definitive treatment for uterine polyps. Misoprostol is a synthetic analogue derived from prostaglandin E1 that has stimulating effects on the smooth muscle fibers of the uterus, causing contractions of the myometrium, which cause endouterine evacuation. The present study shows a possible utility of misoprostol for the conservative treatment of uterine polyps.

ELIGIBILITY:
Inclusion Criteria:

* Women with uterine polyps diagnosed by endovaginal ultrasound and/or hysterosonography, female ≤ 45 years of age

Exclusion Criteria:

* Patients older than 45 years, polyps larger than 60 mm, who did not perform surveillance and/or minimum assessment 6 months after medical management

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Expulsion rate of endometrial polyps | 7 days after misoprostol has been applied

SECONDARY OUTCOMES:
Pregnancy rate after expulsion | 14-21 days after positive β-human Chorionic Gonadotropin (β-hCG)
The pregnancy rate after expulsion in patients with primary sterility | 14-21 days after positive β-hCG

CONTACTS AND LOCATIONS:
Overall Officials: HENRY A MATEO-SÁNEZ, MD, Study Director — Henry Aristoteles Mate-Sánez

IPD SHARING:
Plan to Share IPD: No